CLINICAL TRIAL: NCT05971316
Title: Effectiveness of a Warm-Up With Foam Roller for 3 Months in Professional Basketball Players: A Randomized Controlled Trial
Brief Title: Effectiveness of a Warm-Up With Foam Roller in Professional Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, Javier Reina Abellan, Director, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Universidad Católica de Murcia
Record Dates: First submitted 2023-06-27; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Athletics Injury; Sports Physical Therapy
Keywords: Foam Roller; Performance; Warm-Up; Basketball
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Intervention Model Description: Randomiced Controlled Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Warm-up + Foam Roller (Experimental): General Warm-up + Warm-up with Foam Roller
  Interventions: Device: Foam Roller
- Warm-up Only (No Intervention): General Warm-up only

INTERVENTIONS:
Device: Foam Roller — General Warm-up + Foam Roller
  Arms: Warm-up + Foam Roller

SUMMARY:
The purpose of this study is to analyze the effectiveness of a foam roller warm-up on sports performance in professional basketball players.

DETAILED DESCRIPTION:
Twenty-two professional basketball players, divided into two randomized groups, carried out a specific warm-up for three months with a foam roller. Three measurements were made, pre-intervention, post-intervention at 12 weeks and a four-week follow-up. In these measurements reference data were taken for jumping, ankle dorsiflexion and balance. During this protocol, they performed three series of sixty seconds of application with thirty seconds of rest between series, three days a week and applied to the calf muscles, hamstrings, quadriceps, gluteus and TFL.

ELIGIBILITY:
Inclusion Criteria:

* Masculine or feminine
* Minimum 18 years and maximum 30
* Professional players
* Practice 3 training sessions per week + competition on weekends

Exclusion Criteria:

* Musculoskeletal injury in the last 3 months
* Surgery in the lower extremity in the last year
* Present a diagnosed orthopedic or neurological pathology of the lower limb.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Know the effectiveness of a warm-up with a foam roller in proffesional basketball player during 18 weeks on jumping using the Counter Movement Jump, dorsiflexión using the Lung Test and the balance using the Y-Balance Test | Baseline and week 18
  The countermovement jump will obtain the jump height in centimetres, the ankle dorsiflexion in degrees using the Lung test and the distance in centimeters using the Y-Balance test. High scores in any of the tests will lead to a decrease in the risk of injury and an improvement in performance. A first pre-intervention measurement is carried out, another at 14 weeks post-intervention and others at 18 weeks follow-up. This is the general measure.

SECONDARY OUTCOMES:
Evaluate the improvement obtained in the experimental group after a warm-up protocol with foam roller for 14weeks 3 days per week on the Counter Movement Jump, Lung Test and Y-Balance test vs non-intervention group. | Baseline and week 14
  Observe the differences obtained after 14 weeks between the pre-intervention vs post-intervention measurement in the experimental group and in the control group. This is the specific measure.
Maintenance of foam roller warm-up adaptations on the Counter Movement Jump, Lung Test and Y-Balance Test after intervention for a 1 month | Week 14 and week 18
  To observe if the differences obtained after 14 weeks of intervention are maintained or not during the following 4 weeks of follow-up, between the post-intervention vs. post-follow-up measurement in the experimental group and in the control group. This is a specific measure

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Casado, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- Universidad Católica San Antonio de Murcia, Murcia, Murica, Spain

IPD SHARING:
Plan to Share IPD: No
No research data from the participants is currently shared, the results will be published by the researchers of this study in academic journals. In the future, it is not ruled out making our data and results available to interested researchers and possible collaborators who contact specifically the researchers of our study.

REFERENCES:
- [Derived] Casado D, Nacher I, Pardo J, Reina J. Effectiveness of a Foam Roller Warm-Up in Professional Basketball Players: A Randomized Controlled Trial. Int J Sports Phys Ther. 2025 Jan 1;20(1):15-29. doi: 10.26603/001c.127266. eCollection 2025. PMID 39758693